CLINICAL TRIAL: NCT02808819
Title: A Multicenter, Open-label, Safety Extension Study With Benralizumab (MEDI-563) for Asthmatic Adults on Inhaled Corticosteroid Plus Long-acting β2 Agonist (MELTEMI)
Brief Title: A Safety Extension Study With Benralizumab for Asthmatic Adults on Inhaled Corticosteroid Plus Long-acting β2 Agonist
Acronym: MELTEMI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D3250C00037
Record Dates: First submitted 2016-06-07; First posted 2016-06-22 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Asthma
Keywords: Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Obstructive Lung Diseases
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive | interventions — benralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benralizumab Arm A (Other): Benralizumab administered subcutaneously every 4 weeks
  Interventions: Biological: Benralizumab
- Benralizumab Arm B (Other): Benralizumab administered subcutaneously every 8 weeks
  Interventions: Biological: Benralizumab

INTERVENTIONS:
Biological: Benralizumab — Benralizumab administered subcutaneously every 4 weeks
  Arms: Benralizumab Arm A
Biological: Benralizumab — Benralizumab administered subcutaneously every 8 weeks
  Arms: Benralizumab Arm B

SUMMARY:
The purpose of this study is to continue to characterize the safety profile of benralizumab administration and monitor the pharmacodynamic activity of the drug in those asthma patients who remain on treatment for at least 16 weeks and not more than 40 weeks in the predecessor study D3250C00021 (BORA, NCT02258542).

DETAILED DESCRIPTION:
This is an open-label safety extension study designed to evaluate the safety and tolerability of a fixed 30 mg dose of benralizumab administered subcutaneously (SC) in severe asthma patients on inhaled corticosteroid and long-acting β2 agonist (ICS-LABA) therapy with or without chronic oral corticosteroids (OCS) and/or other asthma controllers. All patients will receive active drug on the same dosing regimen they received in BORA (NCT02258542). In order to protect the blind of BORA, patients will remain blinded to treatment regimen allocation until they have completed all end of treatment (EOT) assessments in BORA and signed informed consent for participation in this study, after which treatment allocation will be unblinded to both the investigator and the patient.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent for study participation must be obtained prior to any study related procedures being performed and according to international guidelines and/or applicable European Union guidelines.
* Female and male patients who have completed at least 16 and not more than 40 weeks in Study D3250C00021.
* Women of childbearing potential (WOCBP) must agree to use an effective form of birth control throughout the study duration and for 16 weeks after the last dose of Investigational Product (IP)
* For WOCBP only: Have a negative urine pregnancy test prior to administration of IP at Visit 1.
* All male patients who are sexually active must agree to use a double barrier method of contraception (condom with spermicide) from the first dose of IP until 16 weeks after their last dose.

Exclusion Criteria:

* Any disorder including but not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric or major physical impairment that is not stable in the opinion of the Investigator and could:

  * Affect the safety of the patient throughout the study
  * Influence the findings of the study or their interpretations
  * Impede the patient's ability to complete the entire duration of study
* A helminth parasitic infection diagnosed during a predecessor study that has either required hospitalization, has not been treated, has been incompletely treated or has failed to respond to standard of care therapy
* Any clinically significant change in physical examination, vital signs, ECG, hematology, clinical chemistry, or urinalysis during the predecessor study which in the opinion of the investigator may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or interfere with the patient's ability to complete the entire duration of the study
* Current malignancy or malignancy that developed during the predecessor study (subjects that had basal cell carcinoma, localized squamous cell carcinoma of the skin which was resected for cure, or in situ carcinoma of the cervix that has been treated/cured will not be excluded).
* Receipt of live attenuated vaccines within 30 days prior to initiation of treatment in this study, during the treatment period, and for 16 weeks (5 half-lives) after the last dose of the IP
* Receipt of immunoglobulin or blood products within 30 days prior to Visit 1
* Planned major surgical procedures during the conduct of the study
* Previous participation in the present study
* Concurrent enrolment in another drug-related interventional clinical trial
* AstraZeneca staff involved in the planning and/or conduct of the study
* Employees of the study center or any other individuals involved with the conduct of the study or immediate family members of such individuals
* Patients with important protocol deviations in the predecessor study at the discretion of the Sponsor
* Patients with ongoing serious adverse events (SAEs) from the prior study should not be enrolled into the this extension study until the SAE has resolved

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-06-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (153):
- United States (45):
  - Research Site, Scottsboro, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Bakersfield, California
  - Research Site, Newport Beach, California
  - Research Site, Redondo Beach, California
  - Research Site, Roseville, California
  - Research Site, Sacramento, California
  - Research Site, San Jose, California
  - Research Site, Stockton, California
  - Research Site, Westminster, California
  - Research Site, Woodland, California
  - Research Site, Colorado Springs, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Doral, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Iowa City, Iowa
  - Research Site, Bangor, Maine
  - Research Site, Quincy, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Traverse City, Michigan
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Jefferson Hills, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Hodges, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, McKinney, Texas
  - Research Site, Abingdon, Virginia
  - Research Site, Falls Church, Virginia
  - Research Site, Madison, Wisconsin
- Argentina (4):
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aire
  - Research Site, La Plata
  - Research Site, Mendoza
- Australia (5):
  - Research Site, Frankston
  - Research Site, Nedlands
  - Research Site, Parkville
  - Research Site, Randwick
  - Research Site, Woolloongabba
- Bulgaria (6):
  - Research Site, Pazardzhik
  - Research Site, Pernik
  - Research Site, Petrich
  - Research Site, Rousse
  - Research Site, Sliven
  - Research Site, Vratsa
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Sherwood Park, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Hamilton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Chile (3):
  - Research Site, Quillota
  - Research Site, Talcahuano
  - Research Site, Valparaíso
- Czechia (4):
  - Research Site, Karlovy Vary
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Rokycany
- France (12):
  - Research Site, Brest
  - Research Site, Dijon
  - Research Site, Le Kremlin-Bicêtre
  - Research Site, Le Mans
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pringy
  - Research Site, Saint-Pierre
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (13):
  - Research Site, Aschaffenburg
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Geesthacht
  - Research Site, Großhansdorf
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Leipzig
  - Research Site, Mainz
  - Research Site, Marburg
  - Research Site, Rüdersdorf
- Poland (26):
  - Research Site, Aleksandrów Łódzki
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Dobre Miasto
  - Research Site, Gdansk
  - Research Site, Gorzów Wlkp
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Kościan
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lubin
  - Research Site, Lublin
  - Research Site, Ostrów Wielkopolski
  - Research Site, Poznan
  - Research Site, Proszowice
  - Research Site, Ruda Śląska
  - Research Site, Rzeszów
  - Research Site, Skierniewice
  - Research Site, Sosnowiec
  - Research Site, Tarnów
  - Research Site, Trzebnica
  - Research Site, Warsaw
  - Research Site, Wieluń
  - Research Site, Wołomin
  - Research Site, Wroclaw
  - Research Site, Żnin
- Russia (7):
  - Research Site, Nizhny Novgorod
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, Vladikavkaz
  - Research Site, Volgograd
  - Research Site, Yekaterinburg
- Spain (5):
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Sagunto(Valencia)
  - Research Site, Salamanca
  - Research Site, Valencia
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Istanbul
- Ukraine (6):
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv Region
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Vinnytsia
- United Kingdom (6):
  - Research Site, Birmingham
  - Research Site, Cambridge
  - Research Site, Chertsey
  - Research Site, Cottingham
  - Research Site, Nottingham
  - Research Site, Stevenage

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSP redacted. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00037&attachmentIdentifier=c52ffe9a-53b4-40d3-935b-1b8ecf80bc07&fileName=d3250c00037-revised-csp-2-redacted.pdf&versionIdentifier=
- See also: SAP redacted. — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00037&attachmentIdentifier=d7b2554d-b014-4ffa-adec-c930fc06f4f5&fileName=d3250c00037-sap-ed-2-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 447 patients enrolled in MELTEMI, 1 patient from Czech Republic was not treated, thus 446 patients received at least 1 dose of IP. Among these treated participants, 347 were from studies SIROCCO(NCT01928771)/CALIMA(NCT01914757) and 99 were from study ZONDA(NCT02075255).
Pre-assignment Details: 170 participants from SIROCCO(NCT01928771)/CALIMA(NCT01914757) assigned to Benralizumab 30 mg every 4 weeks (q4w) with 1 participant not treated. 178 participants from SIROCCO/CALIMA received Benralizumab every 8 weeks (q8w). 51 participants from ZONDA(NCT02075255) received Benralizumab q4w. 48 participants from study ZONDA received Benralizumab q8w.
Groups:
- Benra 30 mg q.4 Weeks: Benralizumab administered subcutaneously every 4 weeks
- Benra 30 mg q.8 Weeks: Benralizumab administered subcutaneously every 8 weeks
Period: Overall Study
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks
Started | 220 | 226
Treated | 220 | 226
Completed | 189 | 195
Not Completed | 31 | 31
Not completed — eg. no treatment efficacy on asthma | 5 | 4
Not completed — Withdrawal by Subject | 10 | 13
Not completed — Site terminated by sponsor | 2 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Lost to Follow-up | 1 | 6
Not completed — Protocol Violation | 0 | 1
Not completed — Development of study-specific withdrawal criteria | 8 | 3
Not completed — Death | 1 | 0
Not completed — Adverse Event | 3 | 4

BASELINE CHARACTERISTICS:
Population: Full analysis set is defined to include subjects who received at least 1 dose of investigational product (IP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 220 | 226 | 446
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (12.00) | 53.0 (11.64) | 53.2 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 144 | 284
  Male | 80 | 82 | 162
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 204 | 206 | 410
  Black or African | 9 | 13 | 22
  American Asian | 5 | 3 | 8
  Other | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Basophils, Full Analysis Set
Description: Change from baseline in hematologic lab parameter of Basophils.
Time Frame: From Week 0 to Benralizumab is available in the local market or early discontinuation. Change from week 0 to the end of treatment period/early discontinuation is presented.
Population: Full analysis set. For each lab test, number of patients is the number of patients with available change from baseline value.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Groups:
- Total: sum per row
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 173 | 178 | 351
10^9 cells/L | 0.014 (0.0229) | 0.012 (0.0243) | 0.013 (0.0236)

2. Primary Outcome: Change From Baseline in Leukocytes, Full Analysis Set
Description: Change from baseline in hematologic lab parameter of Leukocytes.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 178 | 182 | 360
10^9 cells/L | -0.254 (2.0446) | -0.498 (1.7217) | -0.377 (1.8896)

3. Primary Outcome: Change From Baseline in Lymphocytes, Full Analysis Set
Description: Change from baseline in hematologic lab parameter of Lymphocytes.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 173 | 178 | 351
10^9 cells/L | -0.098 (0.5479) | -0.142 (0.6544) | -0.121 (0.6038)

4. Primary Outcome: Change From Baseline in Neutrophils, Full Analysis Set
Description: Change from baseline in hematologic lab parameter of Neutrophils.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 173 | 178 | 351
10^9 cells/L | -0.237 (1.8765) | -0.392 (1.4802) | -0.315 (1.6866)

5. Primary Outcome: Change From Baseline in Monocytes, Full Analysis Set
Description: Change from baseline in hematologic lab parameter of Monocytes.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 173 | 179 | 352
10^9 cells/L | 0.055 (0.1835) | 0.056 (0.1766) | 0.055 (0.1798)

6. Primary Outcome: Change From Baseline in Platelets, Full Analysis Set
Description: Change from baseline in hematologic lab parameter of Platelets.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 177 | 179 | 356
10^9 cells/L | 9.1 (41.72) | 11.9 (36.13) | 10.5 (38.98)

7. Primary Outcome: Change From Baseline in Hematocrit, Full Analysis Set
Description: Change from baseline in hematologic lab parameter of Hematocrit.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: [ratio]
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 172 | 177 | 349
[ratio] | -0.002 (0.0269) | -0.003 (0.0260) | -0.003 (0.0264)

8. Primary Outcome: Change From Baseline in Erythrocytes, Full Analysis Set
Description: Change from baseline in hematologic lab parameter of Erythrocytes.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 178 | 183 | 361
10^12 cells/L | -0.008 (0.2922) | -0.054 (0.2614) | -0.031 (0.2776)

9. Primary Outcome: Change From Baseline in Hemoglobin, Full Analysis Set
Description: Change from baseline in hematologic lab parameter of Hemoglobin.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 178 | 183 | 361
g/L | 2.6 (8.92) | 1.2 (8.37) | 1.9 (8.66)

10. Primary Outcome: Change From Baseline in Alanine Aminotransferase (ALT), Full Analysis Set
Description: Change from baseline in chemistry test ALT.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 174 | 175 | 349
ukat/L | 0.007 (0.2060) | 0.004 (0.2118) | 0.005 (0.2086)

11. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST), Full Analysis Set
Description: Change from baseline in chemistry test AST.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ukat/L
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 174 | 175 | 349
ukat/L | -0.021 (0.1258) | -0.018 (0.1280) | -0.020 (0.1267)

12. Primary Outcome: Change From Baseline in Bilirubin, Full Analysis Set
Description: Change from baseline in chemistry test Bilirubin.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 172 | 175 | 347
umol/L | -0.451 (3.0980) | -0.297 (3.3972) | -0.374 (3.2486)

13. Secondary Outcome: Number of Participants With Asthma Exacerbations During Study Period
Description: Asthma exacerbation is defined by a worsening of asthma requiring the use of systemic corticosteroids for at least 3 days, and/or an in patient hospitalization, and/or an emergency department or urgent care visit
Time Frame: From week 0 to week 184 in study treatment period and through the follow up period (12 weeks from day of last dose). Number and percentage of participants with asthma exacerbation during this period is presented.
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 220 | 226 | 446
Participants | 96 | 97 | 193

14. Secondary Outcome: Number of Participants Who Had Health Care Encounter (ie, Hospitalization, Emergency Department Visits, Urgent Care Visits, and All Other Outpatient Visits Due to Asthma) During Study Period
Description: Hospitalizations, Emergency department (ED) visits, urgent care visits and all other outpatient visits due to asthma
Time Frame: From week 0 to week 184 in study treatment period and through the follow up period (12 weeks from day of last dose). Number and percentage of participants with health care encounters during this period is presented.
Population: Full analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 220 | 226 | 446
Participants | 25 | 28 | 53

15. Secondary Outcome: Change of Blood Eosinophils Count
Description: Change from Baseline to End of Treatment in blood eosinophils count.
Time Frame: as for outcome 1
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: cell/uL
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 173 | 178 | 351
cell/uL | 12.3 (50.24) | -12.9 (212.51) | -0.5 (155.68)

16. Secondary Outcome: Number of Participants With Anti-drug Antibodies (ADA) Responses During the Study
Description: Assessments for the presence of ADA and neutralizing antibody (nAb) throughout study
Time Frame: From week 0 to week 184 in study treatment period and plus 12 weeks follow up period
Population: Full analysis set.
Measure: Number; unit: Participants
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 220 | 226 | 446
Participants
  Positive at any visit: number analyzed (Participants) | 218 | 225 | 443
  Positive at any visit | 19 | 28 | 47
  Both baseline and post-baseline positive: number analyzed (Participants) | 206 | 214 | 420
  Both baseline and post-baseline positive | 11 | 17 | 28
  Only post-baseline positive: number analyzed (Participants) | 211 | 218 | 429
  Only post-baseline positive | 7 | 10 | 17
  ADA Persistently Positive: number analyzed (Participants) | 211 | 218 | 429
  ADA Persistently Positive | 12 | 21 | 33
  ADA Transiently Positive: number analyzed (Participants) | 211 | 218 | 429
  ADA Transiently Positive | 6 | 6 | 12
  Only baseline positive: number analyzed (Participants) | 213 | 221 | 434
  Only baseline positive | 1 | 1 | 2
  nAb positive: number analyzed (Participants) | 218 | 225 | 443
  nAb positive | 13 | 24 | 37
  nAb positive in ADA positive participants: number analyzed (Participants) | 19 | 28 | 47
  nAb positive in ADA positive participants | 13 | 24 | 37

17. Secondary Outcome: Duration of Exposure
Description: Duration of exposure
Time Frame: From week 0 to week 184 in study treatment period
Population: Full analysis set.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks | Total
Number analyzed (Participants) | 220 | 226 | 446
months | 26.35 (10.112) | 25.36 (9.939) | 25.85 (10.026)

ADVERSE EVENTS:
Time Frame: All participants completed treatment period up to Week 184.
Arm/Group | Benra 30 mg q.4 Weeks | Benra 30 mg q.8 Weeks
All-Cause Mortality (participants affected / at risk) | 1/220 | 0/226
Serious Adverse Events (participants affected / at risk) | 44/220 | 47/226
Other Adverse Events (participants affected / at risk) | 169/220 | 145/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg q.4 Weeks (N=220) | Benra 30 mg q.8 Weeks (N=226)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 1 (2)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal stenosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Femoral hernia incarcerated (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Musculoskeletal complication associated with device (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (2) | 0 (0)
Graft infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (4) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood lactic acid increased (Investigations) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bone deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ligament laxity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Silicon granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (2) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 (15) | 13 (19)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Polyarteritis nodosa (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benra 30 mg q.4 Weeks (N=220) | Benra 30 mg q.8 Weeks (N=226)
Diarrhoea (Gastrointestinal disorders) | 8 (12) | 6 (6)
Influenza like illness (General disorders) | 7 (9) | 8 (10)
Acute sinusitis (Infections and infestations) | 13 (20) | 8 (10)
Bronchitis (Infections and infestations) | 23 (33) | 22 (26)
Bronchitis bacterial (Infections and infestations) | 12 (17) | 9 (13)
Influenza (Infections and infestations) | 6 (6) | 10 (10)
Nasopharyngitis (Infections and infestations) | 67 (126) | 64 (112)
Pharyngitis (Infections and infestations) | 10 (19) | 3 (3)
Rhinitis (Infections and infestations) | 11 (18) | 3 (3)
Sinusitis (Infections and infestations) | 17 (26) | 10 (16)
Sinusitis bacterial (Infections and infestations) | 4 (6) | 7 (10)
Upper respiratory tract infection (Infections and infestations) | 14 (20) | 8 (12)
Upper respiratory tract infection bacterial (Infections and infestations) | 10 (19) | 8 (10)
Urinary tract infection (Infections and infestations) | 7 (9) | 7 (7)
Viral upper respiratory tract infection (Infections and infestations) | 29 (38) | 19 (21)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (14) | 10 (10)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 10 (14) | 3 (3)
Dizziness (Nervous system disorders) | 7 (9) | 2 (2)
Headache (Nervous system disorders) | 32 (56) | 21 (41)
Asthma (Respiratory, thoracic and mediastinal disorders) | 16 (21) | 20 (40)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 7 (10) | 4 (4)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 8 (12)
Hypertension (Vascular disorders) | 14 (23) | 24 (31)

LIMITATIONS AND CAVEATS:
All participants in this study had to complete treatment in predecessor studies. Therefore selection bias may exist. Baseline is defined for this study's entry value, not the value prior to Benralizumab treatment. All participants have been treated with Benralizumab prior to this study's entry.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.

DOCUMENTS (2):
  • Study Protocol (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT02808819/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT02808819/SAP_001.pdf